CLINICAL TRIAL: NCT07167888
Title: The Prevalence of Neck and Low Back Pain in Nursing Students at The University of the West Indies, Mona, Jamaica
Brief Title: Low Back and Neck Pain in Nursing Students at The University of The West Indies
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of The West Indies (Other)
Collaborators: The University of The West Indies, Mona (Unknown)
Responsible Party: Principal Investigator, Paula Dawson, MBBS, Head, Physical Medicine and Rehabilitation. Principal Investigator, The University of The West Indies
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CREC-MN.0192,2024/2025
Record Dates: First submitted 2025-09-03; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Back Pain; Low Back Pain; Musculoskeletal Pain; Neck Pain; Spine Health; Musculoskeletal Pain Disorder; Lower Back Pain; Nursing Students; Preclinical Education
Keywords: lower back pain; low back pain; musculoskeletal pain; neck pain; rehabilitation; university student; nursing students; spine health
MeSH Terms: conditions — Back Pain; Low Back Pain; Musculoskeletal Pain; Neck Pain; Collagen Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical Control (Group A) (Experimental): All participants will complete the Cornell Musculoskeletal Discomfort Questionnaires (CMDQ) to assess the frequency, discomfort and interference with work due to musculoskeletal pain; the Numeric Rating Scale (NRS) to assess for perceived pain; as well as Questionnaire A to assess their knowledge, attitude and practice towards musculoskeletal problems of neck or low back pain. Participants who are found to have neck or low back pain will be randomised into two (2) groups: a clinical control group (Group A) and an intervention group (Group B). Group A will not be given any exercise programs over an eight (8) week period after which time, participants will be reassessed using the CMDQ and NRS, as well as a Questionnaire B to evaluate for changes in their knowledge, attitude and practice towards musculoskeletal problems of the neck and low back pain, without having received any intervention.
  Interventions: Behavioral: Clinical Control Group (Group A)
- Spine Exercise Program (Group B) (Experimental): All participants will complete the Cornell Musculoskeletal Discomfort Questionnaires (CMDQ) to assess the frequency, discomfort and interference with work due to musculoskeletal pain; the Numeric Rating Scale (NRS) to assess for perceived pain; as well as Questionnaire A to assess their knowledge, attitude and practice towards musculoskeletal problems of neck or low back pain. Participants who are found to have neck or low back pain will be randomised into two (2) groups: a clinical control group (Group A) and an intervention group (Group B). Group B will be given a standardised spine exercise program over an eight (8) week period, after which time they will be reassessed using the CMDQ and NRS, as well as Questionnaire B to evaluate for changes in their knowledge, attitude and practice towards musculoskeletal problems of the neck and low back pain, having received the intervention.
  Interventions: Behavioral: Spine Exercise Program (Group B)

INTERVENTIONS:
Behavioral: Clinical Control Group (Group A) — The participants who reported the presence of neck or low back pain and were assigned to the clinical control group (Group A) after randomisation will not receive the intervention of an exercise program. The interventional group (Group B) will be asked to keep the standardised exercise program confidential and not share with the control group (Group A). After eight (8) weeks, Group A participants will receive: the Cornell Musculoskeletal Discomfort Questionnaires (CMDQ) to assess for changes in the frequency, discomfort and interference with work due to musculoskeletal pain; a Questionnaire B, to ascertain any changes in their pain level using the Numeric Rating Scale (NRS); as well as their knowledge, attitude and practice towards musculoskeletal problems of the neck and low back pain, without having received any intervention.
  Arms: Clinical Control (Group A)
Behavioral: Spine Exercise Program (Group B) — The standardised spine exercise program will be provided in a handout and given only to the intervention group (Group B), and will include simple basic neck or low back exercises to be done three (3) times per week, as well as brief stretching exercises, to be done during periods of sitting for greater than sixty (60) minutes. The selected participants will be asked to comply with instructions on the handout. Participants who experience worsening of their symptoms, or who develop new symptoms will be assessed as having an adverse outcome and will be withdrawn from the study.
  Arms: Spine Exercise Program (Group B)

SUMMARY:
The purpose of this study is to identify the prevalence of neck and low back pain in nursing students enrolled at the University of the West Indies, Mona; to assess their knowledge, attitude and practice of good spine health and to determine the outcome of a standardised spine exercise program on nursing students experiencing neck and low back pain, using a prospective randomised control design.

DETAILED DESCRIPTION:
Neck and low back pain are among the most common musculoskeletal problems affecting individuals worldwide. Although they are often self-limiting, these conditions may become disabling, significantly impairing productivity, social life, and activities of daily living. Research suggests that approximately 37% of back pain is associated with occupational factors. Prolonged sitting and awkward postures considerably increase the risk of back pain, while neck pain is strongly associated with slouching and repeated or prolonged neck movements. Nursing students, are particularly vulnerable to musculoskeletal pain, and evidence shows that this risk begins as early as their training years. During the preclinical phase of nursing education, students typically spend long hours sitting in lectures, studying, and completing assignments, often with sustained use of computers or tablets. As they progress into their clinical years, nursing students are exposed to a physically demanding environment that involves prolonged standing on ward rounds, assisting during clinical procedures, and performing manual patient handling tasks such as lifting and turning. These activities, when combined with poor ergonomic practices and inadequate core stability, may contribute to the development of neck and low back pain. Alshagga et al. conducted a cross-sectional study in a private Malaysian medical college and reported a higher prevalence of musculoskeletal pain among clinical students, with factors such as increased computer use, elevated BMI, prior trauma, and family history of musculoskeletal disorders playing significant roles. While such studies exist internationally, to the researcher's knowledge, no published study has yet investigated the prevalence of neck and low back pain specifically among nursing students in Jamaica or the wider Caribbean. Exercise therapy is widely recognised as an effective intervention for musculoskeletal pain. Chou and Huffman (2007), in their study on non-pharmacologic therapies for acute and chronic low back pain, demonstrated significant improvements in both pain reduction and function with exercise compared to other noninvasive interventions. Exercise not only strengthens muscles and improves flexibility but also enhances spinal stability and facilitates nutrient transfer to soft tissues, ligaments, and intervertebral discs, thereby promoting spinal health and reducing the risk of injury. The University of the West Indies (UWI), Mona, currently has approximately 400 nursing students enrolled across its four years of training, averaging 130 students per cohort. This study will focus on nursing students enrolled at the UWI Mona to: 1. determine the prevalence of neck and low back pain, 2. assess their knowledge, attitude, and practice toward spine health, and 3. evaluate the effect of a standardised spine exercise program on pain and functional outcomes. Nursing students reporting neck or low back pain will be prospectively randomised into two groups: a control group (Group A) with no intervention, and an intervention group (Group B) that will follow an eight-week standardised spine exercise program. Nursing students will also be assessed to provide a comparative perspective between preclinical and clinical stages of training. Outcome measures will include the Numeric Rating Scale (NRS), the Cornell Musculoskeletal Discomfort Questionnaire (CMDQ), and structured questionnaires designed to evaluate knowledge, attitude, practice, and functional status. To the researcher's knowledge, this will be the first randomised controlled study examining neck and low back pain among nursing students in Jamaica, with the dual aim of establishing prevalence and evaluating the effectiveness of exercise-based intervention strategies in this population. The identity of all participants will be protected and will only be identified by an assigned study number. Basic demographic information, presenting complaints and outcome information will be obtained for the purposes of the study. All data will be managed securely using REDCap, a password-protected, web-based platform compliant with national data protection standards. Data exported for analysis will be handled using SPSS software, ensuring confidentiality is maintained throughout. All records will be securely destroyed three years after study completion.

ELIGIBILITY:
Inclusion Criteria:

1. All students enrolled in the student nursing program at the University of the West Indies, Mona Campus, Jamaica during the period October 4, 2025 to October 3, 2026.
2. Individuals who express a willingness to consent to the study.
3. Individuals who express a willingness to adhere to the standardised exercise program for the stipulated period.

Exclusion Criteria:

1. Individuals with a history of having spine surgery.
2. Individuals who were previously diagnosed with spine pathology and currently receiving rehabilitation therapy.
3. Individuals who express an unwillingness to participate in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Cisgender males and females
Enrollment: 400 (Estimated)
Dates: Start 2025-10-04 (Estimated); Primary Completion 2026-10-03 (Estimated); Study Completion 2026-10-03 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Cornell Musculoskeletal Discomfort Questionnaire (CMDQ) | From enrollment to the end of treatment at eight (8) weeks
  The Cornell Musculoskeletal Discomfort Questionnaire measures the frequency, discomfort and interference with work due to musculoskeletal pain, as reported by participants. The individually reported frequency score is then multiplied by the discomfort score and by the interference score to determine overall severity of pain experienced. This tallied score is then classified by severity into: no discomfort (0), mild (1 to 4.5), moderate (5 to 14), severe (15 - 45) and very severe (45 or higher). All participants will complete this assessment upon enrollment, as well as after an eight (8) week period of treatment, to evaluate any changes in their reported scores.

SECONDARY OUTCOMES:
Knowledge, Attitude and Practice towards Musculoskeletal Problems of Neck and Low back Pain (Questionnaire A) | Done at the time of enrollment (Baseline)
  Questionnaire A is a self-administered general questionnaire used to evaluate knowledge, attitude and practice towards musculoskeletal problems of neck and low back pain.
Change from Baseline in Knowledge, Attitude and Practice Towards Musculoskeletal Problems of Neck and Low Back Pain (Questionnaire B) | From Enrollment to the end of treatment at 8 weeks
  Questionnaire B is a self-administered general questionnaire used to evaluate changes in knowledge, attitude and practice towards musculoskeletal problems of neck and low back pain.
Change from Baseline in the Numeric Rating Scale (NRS) | From Enrollment to the end of treatment at 8 weeks
  The Numeric Rating Scale is a reliable and valid, unidimensional 11-point scale used for patient self-reporting of perceived pain. Its scale uses integers which range from zero (0) to ten (10), where 0 represents no pain, and 10 represents the worst imaginable pain. This is then categorised into mild (1-3), moderate (4-6), and severe (7-10). All participants will complete this assessment upon enrollment, as well as after an eight (8) week period of treatment, to evaluate any changes in their perceived pain. This scale is from public domains and as such, permission for its use is not required.

CONTACTS AND LOCATIONS:
Overall Officials: Paula U.A Dawson, MBBS, Diplomate ABPMR, Principal Investigator — Division of Physical Medicine and Rehabilitation, Faculty of Medical Sciences, The University of the West Indies, Mona, Jamaica.
Locations (1):
- Faculty of Medical Sciences Teaching and Research Complex, University of The West Indies-Mona Campus, Kingston, Jamaica

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] O'Sullivan PB, Phyty GD, Twomey LT, Allison GT. Evaluation of specific stabilizing exercise in the treatment of chronic low back pain with radiologic diagnosis of spondylolysis or spondylolisthesis. Spine (Phila Pa 1976). 1997 Dec 15;22(24):2959-67. doi: 10.1097/00007632-199712150-00020. PMID 9431633
- [Background] Ariens GA, van Mechelen W, Bongers PM, Bouter LM, van der Wal G. Physical risk factors for neck pain. Scand J Work Environ Health. 2000 Feb;26(1):7-19. doi: 10.5271/sjweh.504. PMID 10744172
- [Background] Mandel JH, Lohman W. Low back pain in nurses: the relative importance of medical history, work factors, exercise, and demographics. Res Nurs Health. 1987 Jun;10(3):165-70. doi: 10.1002/nur.4770100308. PMID 2954190
- [Background] Lumbar/Core Strength and Stability Exercise. Athlethic Medicine.
- [Background] Chou R, Huffman LH; American Pain Society; American College of Physicians. Nonpharmacologic therapies for acute and chronic low back pain: a review of the evidence for an American Pain Society/American College of Physicians clinical practice guideline. Ann Intern Med. 2007 Oct 2;147(7):492-504. doi: 10.7326/0003-4819-147-7-200710020-00007. PMID 17909210
- [Background] Smith DR, Leggat PA, Walsh LJ. Workplace hazards among Australian dental students. Aust Dent J. 2009 Jun;54(2):186-8. doi: 10.1111/j.1834-7819.2009.01116_8.x. No abstract available. PMID 19473172
- [Background] Lorusso A, Vimercati L, L'abbate N. Musculoskeletal complaints among Italian X-ray technology students: a cross-sectional questionnaire survey. BMC Res Notes. 2010 Apr 24;3:114. doi: 10.1186/1756-0500-3-114. PMID 20416101
- [Background] Smith DR, Leggat PA. Musculoskeletal disorders among rural Australian nursing students. Aust J Rural Health. 2004 Dec;12(6):241-5. doi: 10.1111/j.1440-1854.2004.00620.x. PMID 15615575
- [Background] Alshagga MA, Nimer AR, Yan LP, Ibrahim IA, Al-Ghamdi SS, Radman Al-Dubai SA. Prevalence and factors associated with neck, shoulder and low back pains among medical students in a Malaysian Medical College. BMC Res Notes. 2013 Jul 1;6:244. doi: 10.1186/1756-0500-6-244. PMID 23815853
- [Background] Solomon A, Wilson S, Meyer M, Sharma N. Prevalence of low back pain among nursing students compared to physical therapy students. International Journal of Nursing Education9(3):115, Jan 2017.
- [Background] Smith DR, Wei N, Ishitake T, Wang RS. Musculoskeletal disorders among Chinese medical students. Kurume Med J. 2005;52(4):139-46. doi: 10.2739/kurumemedj.52.139. PMID 16639985
- [Background] Lis AM, Black KM, Korn H, Nordin M. Association between sitting and occupational LBP. Eur Spine J. 2007 Feb;16(2):283-98. doi: 10.1007/s00586-006-0143-7. Epub 2006 May 31. PMID 16736200
- [Background] Punnett L, Pruss-Utun A, Nelson DI, Fingerhut MA, Leigh J, Tak S, Phillips S. Estimating the global burden of low back pain attributable to combined occupational exposures. Am J Ind Med. 2005 Dec;48(6):459-69. doi: 10.1002/ajim.20232. PMID 16299708
- [Background] Ehrlich GE. Low back pain. Bull World Health Organ. 2003;81(9):671-6. Epub 2003 Nov 14. PMID 14710509
- [Background] Erdinc O HK, Ozkaya M. CROSS-CULTURAL ADAPTATION,VALIDITY AND RELIABILITY OFCORNELL MUSCULOSKELETAL DISCOMFORT QUESTIONNAIRE (CMDQ) IN TURKISH LANGUAGE. 2008.